CLINICAL TRIAL: NCT02397811
Title: Bioavailability Testing of Astaxanthin Formulations
Brief Title: Astaxanthin Formulation Bioavailability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyanotech Corporation (Industry)
Collaborators: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: Pro00019850
Record Dates: First submitted 2015-03-20; First posted 2015-03-25 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-01

CONDITIONS: Bioavailability of Astaxanthin Formulations

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Enteric Coated Softgels (Experimental): Enteric coated softgel capsule containing 4 mg astaxanthin, 3 softgels per dose
  Interventions: Dietary Supplement: Enteric Coated Softgels
- Liposomal Astaxanthin (Experimental): Liposomal astaxanthin containing 4.5 mg astaxanthin per gram. 2.66 grams per dose
  Interventions: Dietary Supplement: Liposomal astaxanthin
- Standard Softgel (Experimental): Standard softgel containing 4 mg per softgel. 3 softgels per dose
  Interventions: Dietary Supplement: Standard Softgel
- Astaxanthin Water Soluble Emulsion (Experimental): Astaxanthin water soluble emulsion containing 1% astaxanthin. 1.2 grams per dose
  Interventions: Dietary Supplement: Astaxanthin Water Soluble Emulsion
- Astaxanthin Water Dispersible Powder (Experimental): Astaxanthin water dispersible powder containing 3% astaxanthin. 0.4 grams per dose
  Interventions: Dietary Supplement: Astaxanthin Water Dispersible Powder
- Standard Softgel with Astaxanthin Gel (Experimental): Statndard softgel with astaxanthin gel containing 4 mg astaxanthin. 3 softgels per dose
  Interventions: Dietary Supplement: Standard Softgel with Astaxanthin Gel

INTERVENTIONS:
Dietary Supplement: Enteric Coated Softgels — Enteric coated softgel capsule containing 4 mg astaxanthin, 3 softgels per dose
  Other Names: BioAstin
  Arms: Enteric Coated Softgels
Dietary Supplement: Liposomal astaxanthin — Liposomal astaxanthin containing 4.5 mg astaxanthin per gram. 3.66 grams per dose
  Other Names: BioAstin
  Arms: Liposomal Astaxanthin
Dietary Supplement: Standard Softgel — Standard softgel containing 4 mg astaxanthin per softgel. 3 softgels per dose
  Other Names: BoAstin
  Arms: Standard Softgel
Dietary Supplement: Astaxanthin Water Soluble Emulsion — Astaxanthin water soluble emulsion containing 1% astaxanthin. 1.2 grams per dose
  Other Names: BioAstin
  Arms: Astaxanthin Water Soluble Emulsion
Dietary Supplement: Astaxanthin Water Dispersible Powder — Astaxanthin water dispersible powder containing 3% astaxanthin. 0.4 grams per dose
  Other Names: BioAstin
  Arms: Astaxanthin Water Dispersible Powder
Dietary Supplement: Standard Softgel with Astaxanthin Gel — Standard softgel with astaxanthin gel containing 4 mg astaxanthin. 3 soft gels per dose
  Other Names: BioAstin
  Arms: Standard Softgel with Astaxanthin Gel

SUMMARY:
Human crossover pharmacokinetic study involving 12 subjects to determine the relative bioavailability of astaxanthin in six commercially available oral formulations.

DETAILED DESCRIPTION:
Astaxanthin is commercially available through several vendors. As a highly-lipophilic compound, its oral bioavailability is likely limited by its solubility in the gut. Pre-formulation strategies for addressing limited solubility include pre-dissolving the astaxanthin in fatty solvents and encapsulating in gelatin capsules. This study will evaluate the oral bioavailability of six different formulations of astaxanthin (12mg) in a double blind crossover study involving 12 subjects.

All subjects will be asked to abstain from consuming any salmon 48hrs before and consuming any food or alcoholic beverages 10 hours before reporting to the blood draw center at 8 AM. They will be fed a standardized breakfast by choosing one of two Jimmy Dean brand breakfast sandwiches (EGG, RED PEPPERS, ONIONS AND PEPPER JACK CHEESE CROISSANT or BACON, EGG & CHEESE BISCUIT. Immediately following the standardized meal, they will take one of six different formulations each containing 12 mg of astaxanthin. Bottled water (Zephyrhills® Brand 100% Natural Spring Water) will be available to each subject ad lib. Blood will be collected immediately before consuming the standardized meal and formulation (0 hr) and then again at 4, 8, 10, and 24 hours post dose by a licensed phlebotomist. In between blood draws, the subjects will be allowed to leave the clinic and allowed to resume their normal diet and lifestyle. However, they will be asked to abstain from consuming any alcoholic beverages or salmon until after completion of the last blood draw at 24hrs. As a measure of quality control, each subject will receive a breathalyzer test for alcohol prior to the 0 and 24 hr blood draws. For each time point, blood will be collected in one 10ml Vacutainer Tube (BD 16x100 containing K2 EDTA) labeled using the randomization scheme to blind the samples. Because 3 of the formulations are powders and the remaining 3 formulations are capsules, which differ slightly size and appearance, neither the subjects nor investigators will be blind to the formulation being tested on any given day. However, each subject will receive separate random assignment to each of the 6 formulations tested over the course of the study and all blood samples will be blinded to the quantitative analysis of astaxanthin plasma levels. This process will be repeated six times for the entire subject population (with-in subject design) with two-week washout periods between each pharmacokinetic (pK) run. The blinded blood samples will be kept refrigerated and will be transported to the Center for Excellence and Brain Repair (CEABR) lab within 24 hours, where it will be processed and subjected to the High pressure liquid chromatograph (HPLC) analysis to quantify the astaxanthin.

ELIGIBILITY:
Inclusion Criteria:Subjects who have signed an informed consent form and who meet all of the following entrance criteria may be enrolled in this clinical trial: Generally healthy men and women who are 21 to 65 years of age, inclusive, at the baseline visit.

-

Exclusion Criteria:Subjects who meet any of the following exclusion criteria are not eligible for participation in this clinical trial:

1. Are unwilling to follow the procedures of the trial, such as making visits or having their blood drawn.
2. Have unintentionally lost or gained 10 or more pounds of body weight in the last 3 months;
3. Have an acute illness (such as a severe cold or flu) or have been hospitalized within the past month for certain conditions;
4. Have severe co-morbid disease including cardiac, pulmonary, renal, hepatic, carotid, peripheral vascular disease, stroke, neurological, clotting disorders or active cancer;
5. Consume alcohol at an elevated level (Defined as consumption of more than 10 standard alcoholic drinks per week. A standard alcoholic drink is defined as one bottle/can of beer (12 ounces) equals one glass of wine (4 ounces) equals one ounce of hard liquor).
6. Have a Body Mass Index (BMI) of less than 15 or greater than 55 m/kg2;
7. Have participated in a clinical trial in the past 4 weeks;
8. Have any disease or condition that in the investigator's opinion compromises the integrity of the clinical trial or the safety of the subject;
9. Severe co-morbid disease is defined as any condition that would cause severe limitations or inability to carry out usual activities of daily living.
10. The exclusion criteria identified above are based upon general safety concerns identified by the study supervisor with input from medical director, or confounders identified by the biostatistician.

    -

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration Cmax) of astaxanthin | 24 hurs
Area under the plasma concentration versus time curve (AUC) of astaxanthin | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- USF Health: College of Medicine, Tampa, Florida, United States

REFERENCES:
- [Background] Baralic I, Djordjevic B, Dikic N, Kotur-Stevuljevic J, Spasic S, Jelic-Ivanovic Z, Radivojevic N, Andjelkovic M, Pejic S. Effect of astaxanthin supplementation on paraoxonase 1 activities and oxidative stress status in young soccer players. Phytother Res. 2013 Oct;27(10):1536-42. doi: 10.1002/ptr.4898. Epub 2012 Nov 28. PMID 23192897
- [Background] Barros MP, Marin DP, Bolin AP, de Cassia Santos Macedo R, Campoio TR, Fineto C Jr, Guerra BA, Polotow TG, Vardaris C, Mattei R, Otton R. Combined astaxanthin and fish oil supplementation improves glutathione-based redox balance in rat plasma and neutrophils. Chem Biol Interact. 2012 Apr 15;197(1):58-67. doi: 10.1016/j.cbi.2012.03.005. Epub 2012 Mar 21. PMID 22465178
- [Background] Bolin AP, Macedo RC, Marin DP, Barros MP, Otton R. Astaxanthin prevents in vitro auto-oxidative injury in human lymphocytes. Cell Biol Toxicol. 2010 Oct;26(5):457-67. doi: 10.1007/s10565-010-9156-4. Epub 2010 Mar 14. PMID 20229275
- [Background] Smith AJ, Kavuru P, Wojtas L, Zaworotko MJ, Shytle RD. Cocrystals of quercetin with improved solubility and oral bioavailability. Mol Pharm. 2011 Oct 3;8(5):1867-76. doi: 10.1021/mp200209j. Epub 2011 Aug 25. PMID 21846121
- [Background] Smith AJ, Kavuru P, Arora KK, Kesani S, Tan J, Zaworotko MJ, Shytle RD. Crystal engineering of green tea epigallocatechin-3-gallate (EGCg) cocrystals and pharmacokinetic modulation in rats. Mol Pharm. 2013 Aug 5;10(8):2948-61. doi: 10.1021/mp4000794. Epub 2013 Jun 26. PMID 23730870